CLINICAL TRIAL: NCT05739864
Title: Evaluation of the Efficacy of Superdonor Fecal Microbiota Transplantation in Patients With Mild-to-moderate Ulcerative Colitis: a Double-blind Randomized Controlled Trial
Brief Title: Superdonor FMT in Patients With Ulcerative Colitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, IANIRO GIANLUCA, Dr., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5184
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Active Ulcerative Colitis
Keywords: Ulcerative Colitis; Fecal Microbiota Trasplantation; Super - donor
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: placebo-controlled, double blind randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To mask treatments to physicisans and recipients, both FMT flasks and syringes will be covered with dark-coloured paper before the infusion, and the patients will be unable to see the endoscopic display during the procedure. Super - donor capsules or placebo ones will look the same. Moreover, the physicians who will evsaluate patients at follow-up will not aware of the treatment being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donor FMT (D-FMT) (Experimental): Patients enrolled in this arm will receive donor FMT
  Interventions: Biological: FMT
- Placebo FMT (P - FMT) (Placebo Comparator): Patients enrolled in this arm will receive placebo FMT
  Interventions: Other: Placebo FMT

INTERVENTIONS:
Biological: FMT — This intervention is represented by the administration, in the recipients' gut, of super - donor microbiota through FMT
  Arms: Donor FMT (D-FMT)
Other: Placebo FMT — This intervention is represented by the administration, in the recipients' gut, of a placebo through FMT
  Arms: Placebo FMT (P - FMT)

SUMMARY:
In the last decades fecal microbiota transplantation (FMT) has been established as a highly effective option in the treatment of recurrent Clostridioides difficile infection (rCDI), with a success rate of nearly 90%. For this reason, it is recommended by international guidelines as a treatment option for this indication in clinical practice.

Recently, a considerable body of evidences, suggest FMT as an effective and safe treatment in patients affected by Ulcerative Colitis (UC). In a recent meta-analysis of 324 subjects with UC, 30.4% of patients achieved both clinical and endoscopic remission after FMT compared to placebo (9.8%, P<0.00001). However, among the various published trials there is a fair variability in terms of methods and results, which are not comparable to those obtained in the rCDI.

Nowadays, one of the most critical factors involved in the effectiveness of FMT in UC patients, is the choice of the donor.

In addition, several studies have shown that some donors are associated with a higher clinical response rate than others. This hypothesis has been demonstrated in patients affected by irritable bowel syndrome, in which the use of a super-donor (a healthy person who has the predictive clinical and lifestyle characteristics of a healthy microbiota, and with a microbial profile associated with favorable clinical conditions) resulted in significantly higher clinical efficacy rates than placebo, similar to those obtained in rCDI (89%).

Currently, studies that explored the efficacy of the super-donor FMT in UC patients are not yet available. Aim of this study is to investigate the efficacy of super - donor FMT, compared with placebo FMT, in the treatment of UC. The investigators will randomize adult patients with a recent diagnosis of UC to FMT from super - donors or placebo, by colonoscopy (first infusion) and capsules administration. Then, patients will be followed up 2 months after FMT.

DETAILED DESCRIPTION:
In the last decades fecal microbiota transplantation (FMT) has been established as a highly effective option recurrent Clostridioides difficile infection (rCDI) treatment, with a success rate of nearly 90%. For this reason, it is recommended by international guidelines as a treatment option for this indication in clinical practice.

Recently, a considerable body of evidence supports FMT as an effective and safe treatment in patients affected by Ulcerative Colitis (UC). In a recent meta-analysis of 324 subjects with UC, 30.4% of patients achieved both clinical and endoscopic remission after FMT compared to placebo (9.8%, P<0.00001). However, among the various published trials there is a fair variability in terms of methods and results, which are not comparable to those obtained in the rCDI.

Nowadays, one of the most critical factors involved in the effectiveness of FMT in UC patients is the choice of the donor. In addition, several studies have shown that some donors have been associated with a higher clinical response rate than others. This hypothesis has been demonstrated in patients affected by irritable bowel syndrome, in which the use of a super-donor (a healthy person who has the predictive clinical and lifestyle characteristics of a healthy microbiota, and with a microbial profile associated with favorable clinical conditions) resulted in significantly higher clinical efficacy rates than placebo, similar to those obtained in rCDI (89%).

Currently, studies that explored the efficacy of the superdonor FMT in UC patients are not yet available.

The extended aims of this study are:

* To compare the efficacy of superdonor FMT and placebo FMT in treating mild-to-moderate Ulcerative Colitis.
* To investigate changes in gut microbiome after treatments
* To investigate changes in serum cytokines after treatments
* To investigate changes in disease activity, investigated by the use of partial mayo score, after treatments.

The investigators will carry out a single-centre double blind, placebo-controlled, randomized clinical trial of super - donor FMT vs placebo FMT in patients with mild-to-moderate UC Patients will be recruited among those referred to the gastroenterology unit of the Fondazione Policlinico Universitario "A. Gemelli". Patients with all inclusion criteria and none of the exclusion criteria (detailed in the specific section of this website) will be considered for this study.

Before randomization, demographic data will be collected by the gastroenterology staff.

Moreover, patients will be requested to give stool samples to be collected in a sterile, sealed container and stored at -80°C for metagenomic assessment of gut microbiome by the microbiology staff. Additionally, a blood sample will be collect for cytokine immunoassays.

After baseline assessments, patients will be randomly assigned to one of the following treatment arms:

* Donor FMT (D-FMT)
* Placebo FMT (P-FMT) Patients in both groups will undergo three FMT procedure. Each patient in the D-FMT group will receive feces from one single donor. Placebo FMT will be made of 250 mL water for colonoscopy or using empty capsules. The selection of stool donors will be performed by the gastroenterology staff following protocols previously recommended by international guidelines and according the new recommendation imposed by the reorganization of fecal microbiota transplant during the COVID-19 pandemic. The assignment of fecal infusates from healthy donors to patients will be done randomly, without any specific recipient-donor match, as this is not recommended by international guidelines All fecal infusates and capsules will be manufactured in the microbiology unit of our hospital. Only frozen feces will be used. Preparation of frozen feces will follow protocols from international guidelines. Patients in both groups will undergo the first infusion by colonoscopy. Then, patients will receive frozen fecal capsules ( 15 capsules b.i.d.) at 3 and 7 days after the first FMT.

Furthermore, patients in the D-FMT group receive a pre-conditioning with vancomycin and neomycin+bacitracin for 3 days, because published data from our group show that pre-FMT antibiotics are associated with higher rates of microbial engraftment rates and increased clinical response regardless of the disease.

Patients of the P-FMT group will receive a pre-conditioning with placebo at the same dose.

Follow-up visits will be performed by physicians from the gastroenterology unit. All patients will be followed up for 2 months after the end of treatments. Follow-up visits will be scheduled at week 1, week 4, and week 8, after the end of treatments.

At each visit the following assessments will be performed: 1) collection of stool samples for microbiome analysis; 2) collection of blood sample for cytokine immunoassay; 3) record of adverse events. Unscheduled follow-up visits will be offered if requested by the patients.

Study Outcomes are detailed in the specific section of this website. The statistical analysis will be performed both on an intention-to-treat and per-protocol basis. Differences among groups will be assessed with a two tailed Wilcoxon-rank sum test for continuous data and with Fisher's exact probability test (using two-tailed P-values) for categorical data. Differences in cure percentages will be determined with Fisher's exact test (with two-tailed P values). Microbiome analysis will be performed with shotgun sequencing techniques. For microbiome analysis statistical differences between group means will be calculated using a two-tailed Wilcoxon-Rank Sum Test, through the R statistical software package (R Core Team, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old
* Mild to Moderate Ulcerative Colitis (total Mayo score 3 -10 + endoscopic subscore ≥ 1) in stable maintenance therapies (> 4 weeks with Aminosalicylates, > 6 weeks with immunosuppressant or biologics agents);
* Recent diagnosis (< 12 months) of Ulcerative Colitis;
* Ability to provide written informed consent
* Ability to be compliant with the scheduled procedures

Exclusion Criteria:

* Age < 18 years old
* Known active gastrointestinal disorders (e.g. infectious gastroenteritis, coeliac disease, Crohn disease, irritable bowel syndrome, chronic pancreatitis, biliary salt diarrhoea)
* Previous colorectal surgery or cutaneous stoma
* Current or recent (< 2 weeks) therapy with drugs that could possibly alter gut microbiota (e.g. antimicrobials, probiotics, proton pump inhibitors or metformin)
* Decompensated heart failure or heart disease with ejection fraction lower than 30%
* Severe respiratory insufficiency
* Psychiatric disorders
* Pregnancy or breastfeeding
* Unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Number of patients who will obtain remission of disease 8 weeks after treatments | 2 months
  The investigators will evaluate evaluate the number of participants who will obtain disease remission (assessed by total mayo score </= 2, or endoscopic Mayo </= 1) 8 weeks after treatments.

SECONDARY OUTCOMES:
Number of patients who will obtain remission of disease 1 and 4 weeks after treatments. | 1 months
  The investigators will evaluate evaluate the number of participants who will obtain disease remission (assessed by total mayo score </= 2, or endoscopic Mayo </= 1) 1 and 4 weeks after treatments.
Number of patients who will obtain clinical disease remission 1,4 and 8 weeks after treatments. | 2 months
  The investigators will evaluate the number of participants who will obtain clinical disease remission (SSCAI score ≤2) 1,4 and 8 weeks after treatments.
Number of patients who will obtain endoscopic remission 1,4 and 8 weeks after treatments | 2 months
  The investigators will evaluate the number of participants who will obtain endoscopic remission (endoscopic Mayo score <1) 1,4 and 8 weeks after treatments
Number of patients who will obtain clinical response | 2 months
  The investigators will evaluate the number of participants who will obtain clinical response, defined as a reduction ≥ 3 points of total Mayo score, 1,4 and 8 weeks after treatments.
Evaluation of changes in recipients' microbiome after treatments, at each time point. | 2 months
  The investigators will evaluate the characteristics of recipients' microbiome, assessed by metagenomics analysis, 1,4 and 8 weeks days after treatments, compared to baseline and super - donors' microbiome.
Evaluation of changes in serum cytokines after treatments, at each time point. | 2 months
  The investigators will evaluate the characteristics of patients serum cytokines, 1,4 and 8 weeks days after treatments compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Ianiro, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Gianluca Ianiro, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other researchers
Supporting Information: Study Protocol
Time Frame: data will be available after the completion of the study, for 5 years
Access Criteria: Data will be given upon request to the PI